CLINICAL TRIAL: NCT01313559
Title: An Open Label Randomized Phase II Study of SOM230 and Everolimus in Castrate-Resistant, Chemotherapy-Naïve Prostate Cancer Patients
Brief Title: Pasireotide (SOM230) With or Without Everolimus in Treating Patients With Hormone Resistant, Chemotherapy Naive Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11D.78; 2010-52 (Other: CCRRC); JT 2184 (Other: JeffTrial Number)
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Results first posted 2018-01-16 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Castrate Resistant Prostate Cancer; Chemotherapy Naive Prostate Cancer; Prostate Cancer
Keywords: Castrate Resistant; Chemotherapy Naive; Prostate Cancer; SOM230; Everolimus
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pasireotide; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A (pasireotide) (Active Comparator): Patients receive pasireotide IM once every 4 weeks
  Interventions: Drug: Pasireotide; Other: Laboratory biomarker analysis
- Cohort B (pasireotide and everolimus) (Experimental): Patients receive pasireotide as in cohort A and everolimus PO QD
  Interventions: Drug: Pasireotide; Drug: Everolimus; Other: Laboratory biomarker analysis

INTERVENTIONS:
Drug: Pasireotide — Given IM
  Other Names: SOM230
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001
  Arms: Cohort B (pasireotide and everolimus)
Other: Laboratory biomarker analysis — Correlative studies

SUMMARY:
This is an open label randomized phase II study for prostate cancer patients who have disease progression after hormonal therapy. SOM230 LAR (Pasireotide) binds to its receptor of prostate cancer cells and can prevent them from growing. Everolimus works by targeting a cell survival factor in prostate cancer. The combination of these drugs may work better for the treatment of prostate cancer without toxic chemotherapy. Patients will receive either SOM230 LAR (group A) or SOM230 LAR in combination with Everolimus (group B).

DETAILED DESCRIPTION:
Prostate cancer cells typically have neuroendocrine (NE) differentiation features after they become resistant to hormonal therapy. Somatostatin (SST - a peptide hormone) receptors (SSTR) are usually expressed in a high level in these advanced prostate cancer cells. When SSTR is activated pharmacologically by drugs similar to SST, prostate cancer cell growth is inhibited. SOM230 is a new agent which can activate SSTR and block other key survival molecules/pathways such as phosphatidylinositol 3-kinases (PI3K), mitogen-activated protein (MAP) kinases (MAPK) signaling pathways. Thus SOM230 itself has anticancer activity for prostate cancer.

It is also well known that hormonal refractory prostate cancer can grow in an environment of very low male hormone level because of the activation of several non-androgen receptor survival pathways. One key survival pathway is mediated by an important molecule called mammalian target of rapamycin (mTOR). Drugs, such as Everolimus, have anticancer activity in prostate cancer pre-clinically, but do not sustain its activity. The reason was that cancer cells can up-regulate other survival pathways such as PI3K, MAPK, thus bypass mTOR.

It is hypothesized that SOM230 not only have anti-tumor effect in prostate cancer directly, but also can block the up-regulated (feed-back loop), alternative PI3K or MAPK survival pathways induced by mTOR inhibitors.

The goal of this study is to develop a new well tolerated therapy that can be offered to prostate cancer patients prior to receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age minimum: 18 years old
* Histological confirmation of prostatic adenocarcinoma
* PSA > or = to 2 ng/ml
* PSA progression (serially rises on two occasions each at least one week apart) OR disease progression on imaging studies (CT scan or bone scan).
* Minimally symptomatic - no symptoms attributed to prostate cancer greater than Grade I based on NCI CTCAE Version 4.0 grading of toxicities
* Discontinuation of all antiandrogen, ketoconazole and investigational drugs for at least 4 weeks (6 weeks for bicalutamide) prior to study initiation
* Maintain castrate levels of testosterone (<50ng/dL)
* Karnofsky Performance Status > or = to 60%
* Life expectancy > 3 months
* Adequate hematologic, renal, and liver function

Exclusion Criteria:

* Currently active second malignancy other than non-melanoma skin cancers.
* Clinically significant cardiovascular disease: EF < 30%, NHYA Class III or greater congestive heart failure, myocardial infarction/unstable angina within 6 months prior to study enrollment, or significant ECG abnormalities such as QRS/QT prolongation (see Section 5.3).
* Progressive pulmonary disease, such as advanced COPD, pulmonary fibrosis, or supplemental O2 requirement.
* Known CNS disease, except for treated brain metastases.
* Poorly controlled diabetes mellitus (HbA1c > 7 %) or fasting blood glucose level >126 mg/dL in non-diabetic patients or > 189 mg/dL in diabetic patients (can be enrolled after initiation or titration of anti-diabetic agent(s)).
* Poorly controlled hypercholesterolemia (fasting serum cholesterol >300 mg/dL) or hypertriglyceridemia (> 2.5 x ULN). Patients above either threshold can be included after initiation of appropriate lipid lowering medication.
* Current use of chronic steroids (equivalent of 20mg prednisone daily). Inhaled steroids are acceptable.
* Active gallbladder disease or hepatitis (AST or ALT > 2.0, or bilirubin > 1.5x ULN), liver cirrhosis, or severe liver impairment (Child-Pugh class C). It is highly recommended that patients positive for HBV-DNA or HBsAg are treated prophylactically with an antiviral for 1-2 weeks prior to receiving study drug.
* Serum creatinine >1.5 upper limit of normal or on dialysis.
* Prior use of a somatostatin analog or mTOR inhibitor for the treatment of PC.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09-15 (Actual); Study Completion 2012-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianqing Lin, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (2):
- United States (2):
  - Yale Cancer Center, New Haven, Connecticut
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A (Pasireotide) | Cohort B (Pasireotide and Everolimus)
Started | 4 | 2
Completed | 0 | 0
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Disease progression | 1 | 0
Not completed — Rising PSA | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Pasireotide) | Cohort B (Pasireotide and Everolimus) | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 4 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.0 (4.6) | 69.4 (8.4) | 75.2 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Alive and Progression Free After 12 Weeks of Treatment
Description: Progression of disease is defined as disease progression by RECIST 1.1 criteria on CT scan (X-ray computed tomography), or appearance of > 2 new bone lesions on bone scan, or prostate-specific antigen (PSA) progression by Prostate Cancer Clinical Trials Working Group (PCWG2) criteria or death from any cause.
Time Frame: 12 weeks after treatment
Measure: Number; unit: participants
Arm/Group | Cohort A (Pasireotide) | Cohort B (Pasireotide and Everolimus)
Number analyzed (Participants) | 4 | 2
participants | 0 | 0

2. Secondary Outcome: Number of Participants With > 50% Decline From Baseline PSA Level
Time Frame: After 12 weeks of treatment
Measure: Number; unit: participants
Arm/Group | Cohort A (Pasireotide) | Cohort B (Pasireotide and Everolimus)
Number analyzed (Participants) | 4 | 2
participants | 2 | 0

3. Secondary Outcome: Number of Participants Without New Bone Lesions After 12 Weeks of Treatment
Time Frame: After 12 weeks of treatment
Measure: Number; unit: participants
Arm/Group | Cohort A (Pasireotide) | Cohort B (Pasireotide and Everolimus)
Number analyzed (Participants) | 4 | 2
participants | 0 | 0

4. Secondary Outcome: Number of Participants With Progression Free Survival (PFS) Based on RECIST 1.1 Criteria
Description: Progression free survival (PFS) based on primary outcome criteria for disease progression. Patients without radiographic disease progression who permanently discontinue the study drugs will be censored
Time Frame: Assessed up to 30 days after completion of study treatment
Measure: Number; unit: participants
Arm/Group | Cohort A (Pasireotide) | Cohort B (Pasireotide and Everolimus)
Number analyzed (Participants) | 4 | 2
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Cohort A (Pasireotide) | Cohort B (Pasireotide and Everolimus)
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/2
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Pasireotide) (N=4) | Cohort B (Pasireotide and Everolimus) (N=2)
Elevated creatinine (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Pasireotide) (N=4) | Cohort B (Pasireotide and Everolimus) (N=2)
Abdominal pain (General disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anorexia (General disorders) | 2 (2) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cough (General disorders) | 1 (1) | 1 (1)
Decreased appetite (General disorders) | 0 (0) | 1 (1)
Dehydration (General disorders) | 2 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (2)
Dizziness (General disorders) | 2 (3) | 0 (0)
Dry mouth (General disorders) | 1 (1) | 1 (1)
Dry skin (General disorders) | 0 (0) | 1 (1)
Dysgeusia (General disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Elevated creatinine (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Elevated transaminase (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fall (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (4)
Flatulence (General disorders) | 2 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 3 (4) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hip pain (General disorders) | 0 (0) | 1 (1)
Hot flashes (General disorders) | 1 (1) | 0 (0)
Hyperglycemia (Blood and lymphatic system disorders) | 3 (5) | 2 (6)
Hypertension (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypocalcemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Mood alteration (General disorders) | 1 (1) | 0 (0)
Mucositis (General disorders) | 0 (0) | 2 (2)
Muscular pain (General disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 1 (1) | 0 (0)
Pain at injection site (General disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Shoulder pain (General disorders) | 0 (0) | 1 (1)
Side pain (General disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sweating (General disorders) | 0 (0) | 2 (2)
Tremors (General disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (General disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Vomiting (General disorders) | 1 (1) | 1 (1)
Weakness (General disorders) | 1 (1) | 0 (0)
Weight loss (General disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Study terminated prematurely due to slow accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes